CLINICAL TRIAL: NCT04070131
Title: Rehabilitació Assistida Amb Cavalls Posttractament oncològic en Nens i Adolescents: Efectes físics i psicològics
Brief Title: Horse Assisted Rehabilitation Postoncologic Treatment in Children and Adolescents: Physical and Psychological Effects
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Escoles Universitaries Gimbernat (Other)
Collaborators: Hospital Vall d'Hebron (Other); Hospital Sant Joan de Deu (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HARHB
Record Dates: First submitted 2019-08-21; First posted 2019-08-28 (Actual); Last update posted 2022-03-23 (Actual); Status verified 2022-03

CONDITIONS: Cancer; Child, Only; Child Behavior; Neurologic Gait Disorder; Neurologic Complication
Keywords: Child Behavior; Neurologic Gait Disorder; Cancer; Physical Therapy Modalities; Physical Therapy Specialty; Physical and Rehabilitation Medicine; Rehabilitation
MeSH Terms: conditions — Neoplasms; Child Behavior; Gait Disorders, Neurologic | interventions — Equine-Assisted Therapy

STUDY DESIGN:
Intervention Model Description: Controlled parallel clinical trial, randomised, not-masked, with Control Group and Intervention Group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (No Intervention): Regular follow ups.
- Intervention Group (Experimental): One weekly session (1 hour) of Horse-Assisted Rehabilitation, 24 weeks.
  Interventions: Other: Horse-Assisted Rehabilitation

INTERVENTIONS:
Other: Horse-Assisted Rehabilitation — One hour weelky session of hippotherapy.
  Other Names: Equine-Assisted Rehabilitation; Hippotherapy
  Arms: Intervention Group

SUMMARY:
Clinical trial on the physical and psychological effects of Horse Assisted Rehabilitation after the treatment of cancer in children 4 to 18 years of age.

DETAILED DESCRIPTION:
Randomized controlled open labelled trial. Duration: 6 months. Groups: Control Group (standard follow-up) and Intervention Group (one weekly rehabilitation session assisted by horse). Participants: 30 children, 4 to 18 years of age, after 6 months of the discharge of the cancer treatment with nervous system involvement.

ELIGIBILITY:
Inclusion Criteria:

* Children between 4 and 18 years of age, who had suffered a cancer with affectation of the Central Nervous System
* With or without motor, functional and / or cognitive deficits or neurological disorders due to their basic problem or be as a consequence of the therapeutic procedures, with any degree of disability
* More than 6 months after receiving the discharge of oncology (chemotherapy or radiotherapy)

Exclusion Criteria:

* Immunodepression
* Hypotonia with severe pelvic instability that does not allow seating on the horse safely
* Weight greater than 80Kg.
* Phobia to horses

Ages: 4 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 2019-10-15 (Actual); Primary Completion 2022-02-01 (Actual); Study Completion 2022-06-01 (Estimated)

PRIMARY OUTCOMES:
Self-Reported Quality Of Life Changes | Baseline and 25th week
  Pediatric Quality of Life Inventory - Child-Self Report (PedsQL-C) (PedsQL is a model for measuring quality of life in children with acute or chronic pathology; The PedsQL questionnaire is composed of 23 items comprising 4 dimensions; items are reversed scored and linearly transformed to a 0-100 scale; in order to get a total score we must sum all the items scores over the number of items answered on all the Scales; total score 0-100, higher=better).

SECONDARY OUTCOMES:
Parent-Proxys Reported Quality Of Life Changes | Baseline and 25th week
  Pediatric Quality of Life Inventory - Parent-Proxy Report (PedsQL-PC) (PedsQL is a model for measuring quality of life in children with acute or chronic pathology; The PedsQL questionnaire is composed of 23 items comprising 4 dimensions; items are reversed scored and linearly transformed to a 0-100 scale; in order to get a total score we must sum all the items scores over the number of items answered on all the Scales; total score 0-100, higher=better).
General Health Status Changes | Baseline and 25th week
  Barcelona General Health Status Questionnaire 2000 (sections: C, D, E, F, K, L, M; qualitative questionnaire, no total score).
Anxiety Changes | Baseline and 25th week
  State Trait Ansiety IInventory for children (STAI-CH) - norm-referenced scores (T scores and percentile ranks) for each one of the two subscales: Anxiety-Trait & Anxiety-State (scores 0-60 in each subscale, higher = worse).
Depression Changes | Baseline and 25th week
  Childhood Depression Inventory (CDI), self report long version (28 items) to assess the presence and severity of depressive symptoms in children. Scores range from 0-56, with higher scores indicating higher levels of depression.
Behavior Changes | Baseline and 25th week
  Behavior Assessment System for Children - Parent Rating Scale (BASC-PRS), second version (BASC-2) - BASC-2 is parent-reported, well-established scale for externalizing/internalizing problem of children and adolescents. Scoring manual and software is provided by the assessment developers; norm-referenced scores (T scores and percentile ranks) are available in the score reports, as are interpretations of strengths and weaknesses and target behaviors for intervention (mean of 50 and standard deviation of 10; for the behavior problem scales, scores above 60 are considered problematic; for the adaptive scales, scores below 40 are considered problematic).
Self-Reported Physical Function Changes | Baseline and 25th week
  PedsQL-C (subscale Health and Activities: to create Scale Scores, the mean is computed as the sum of the items over the number of items answered; next, sum the item scores and divide by the number of items in the scale minus Nmiss)
Parents-Reported Physical Function Changes | Baseline and 25th week
  PedsQL-PC (subscale Physical Functioning: to create Scale Scores, the mean is computed as the sum of the items over the number of items answered; next, sum the item scores and divide by the number of items in the scale minus Nmiss)
Self-Reported Emotional Function Changes | Baseline and 25th week
  PedsQL-C (subscale Feelings: to create Scale Scores, the mean is computed as the sum of the items over the number of items answered; next, sum the item scores and divide by the number of items in the scale minus Nmiss)
Parent-Reported Emotional Function Changes | Baseline and 25th week
  PedsQL-PC (subscale Emotional Functioning: to create Scale Scores, the mean is computed as the sum of the items over the number of items answered; next, sum the item scores and divide by the number of items in the scale minus Nmiss)
Self-Reported Sociability Function Changes | Baseline and 25th week
  PedsQL-C (subscale Get Along with Others: to create Scale Scores, the mean is computed as the sum of the items over the number of items answered; next, sum the item scores and divide by the number of items in the scale minus Nmiss)
Parent-Reported Sociability Function Changes | Baseline and 25th week
  PedsQL-PC (subscale Emotional Functioning: to create Scale Scores, the mean is computed as the sum of the items over the number of items answered; next, sum the item scores and divide by the number of items in the scale minus Nmiss)
Balance Changes | Baseline, 6th, 12th and 25th week
  Pediatric Balance Scale (PBS: 14-item, criterion-referenced measure, which examines functional balance in the context of everyday tasks; Scoring (0-4) is based on how long a specific movement or position is performed, how long the position can be maintained, or how much assistance it requires. The highest score in PBS is 56, higher is better).
Position Changes | Baseline, 6th, 12th and 25th week
  Sitting Assessment Scale (Sitting Assessment Scale (SAS) is a standardized observational instrument designed for assessment of sitting in children with cerebral palsy (CP); the scale is composed of five items evaluating head, trunk and foot control and arm and hand function, where each item is assessed with a score from 1 to 4 (1 =none; 2=poor; 3=fair; 4=good) and each score (1,2,3,4) has specific decriptors of each item of the SAS).
Proprioception-Coordination Changes | Baseline and 25th week
  Developmental Coordination Disorder Questionnaire 2007 (DCDQ'07: the DCDQ is a brief questionnaire designed to screen for coordination disorders in children, aged 5 to 15 years, and consists of 15 items grouped into three distinct factors (motor control during movement, fine motor and handwriting and general coordination; to reach scores, sum each column to compute the numbers onto the Score Sheet, and add all factor scores to compute a Total Score: 0-75, higher is better).
Autonomous Neurvous System activation function Changes | Baseline, 6th, 12th and 25th week
  Heart Rate Variability (HRV, low/high frequency (LH/FH) power ratio; modulation of heart rate variability assessed through analysis of data collected by HRV wireless monitorisation and PolarH7(R) thoracic band (medical device), following the American and European Cardiological Societies).

CONTACTS AND LOCATIONS:
Overall Officials: Jordi Esquirol Caussa, PhD, MD, Study Director — Escoles Universitàries Gimbernat; Teresa Xipell Prunés, PT, Principal Investigator — Escoles Universitàries Gimbernat
Locations (2):
- Spain (2):
  - Hospital Universitari de Sant Joan de Déu, Esplugues de Llobregat, Barcelona
  - Hospital Universitari Vall d'Hebron, Barcelona

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Signorelli C, Wakefield CE, Fardell JE, Wallace WHB, Robertson EG, McLoone JK, Cohn RJ. The impact of long-term follow-up care for childhood cancer survivors: A systematic review. Crit Rev Oncol Hematol. 2017 Jun;114:131-138. doi: 10.1016/j.critrevonc.2017.04.007. Epub 2017 Apr 13. PMID 28477741
- [Background] Miller K, Mehta R, Abraham J, Opneja A, Jain RK. Patterns of Long-term Cancer Survivorship Care in a National Cancer Institute-Designated Comprehensive Cancer Center. Am J Clin Oncol. 2017 Dec;40(6):639-643. doi: 10.1097/COC.0000000000000217. PMID 26359697
- [Background] Ford JS, Chou JF, Sklar CA. Attendance at a survivorship clinic: impact on knowledge and psychosocial adjustment. J Cancer Surviv. 2013 Dec;7(4):535-43. doi: 10.1007/s11764-013-0291-9. Epub 2013 Jun 22. PMID 23793467
- [Background] Hooke MC, Gilchrist L, Foster L, Langevin M, Lee J. Yoga for Children and Adolescents After Completing Cancer Treatment. J Pediatr Oncol Nurs. 2016 Jan-Feb;33(1):64-73. doi: 10.1177/1043454214563936. Epub 2015 Feb 2. PMID 25643973
- [Background] Rigby BR, Grandjean PW. The Efficacy of Equine-Assisted Activities and Therapies on Improving Physical Function. J Altern Complement Med. 2016 Jan;22(1):9-24. doi: 10.1089/acm.2015.0171. Epub 2015 Dec 14. PMID 26654868
- [Background] Hilliere C, Collado-Mateo D, Villafaina S, Duque-Fonseca P, Parraca JA. Benefits of Hippotherapy and Horse Riding Simulation Exercise on Healthy Older Adults: A Systematic Review. PM R. 2018 Oct;10(10):1062-1072. doi: 10.1016/j.pmrj.2018.03.019. Epub 2018 Apr 5. PMID 29626616
- [Background] Koca TT, Ataseven H. What is hippotherapy? The indications and effectiveness of hippotherapy. North Clin Istanb. 2016 Jan 15;2(3):247-252. doi: 10.14744/nci.2016.71601. eCollection 2015. PMID 28058377
- [Background] Cerulli C, Minganti C, De Santis C, Tranchita E, Quaranta F, Parisi A. Therapeutic horseback riding in breast cancer survivors: a pilot study. J Altern Complement Med. 2014 Aug;20(8):623-9. doi: 10.1089/acm.2014.0061. Epub 2014 Jun 25. PMID 24963599
- [Background] Lee PT, Dakin E, McLure M. Narrative synthesis of equine-assisted psychotherapy literature: Current knowledge and future research directions. Health Soc Care Community. 2016 May;24(3):225-46. doi: 10.1111/hsc.12201. Epub 2015 Mar 2. PMID 25727575
- [Background] Kang KD, Jung TW, Park IH, Han DH. Effects of Equine-Assisted Activities and Therapies on the Affective Network of Adolescents with Internet Gaming Disorder. J Altern Complement Med. 2018 Aug;24(8):841-849. doi: 10.1089/acm.2017.0416. Epub 2018 Apr 26. PMID 29698054
- [Background] Pendry P, Carr AM, Smith AN, Roeter SM. Improving adolescent social competence and behavior: a randomized trial of an 11-week equine facilitated learning prevention program. J Prim Prev. 2014 Aug;35(4):281-93. doi: 10.1007/s10935-014-0350-7. PMID 24898318
- [Background] Garner BA, Rigby BR. Human pelvis motions when walking and when riding a therapeutic horse. Hum Mov Sci. 2015 Feb;39:121-37. doi: 10.1016/j.humov.2014.06.011. Epub 2014 Nov 28. PMID 25436916
- [Background] Fazio E, Medica P, Cravana C, Ferlazzo A. Hypothalamic-pituitary-adrenal axis responses of horses to therapeutic riding program: effects of different riders. Physiol Behav. 2013 Jun 13;118:138-43. doi: 10.1016/j.physbeh.2013.05.009. Epub 2013 May 15. PMID 23684906
- [Background] Herrero Gallego P, García Antón E, Monserrat Cantera ME, Oliván Blázquez B, Gómez Trullén EM, Trenado Molina J. Efectos terapéuticos de la hipoterapia en la parálisis cerebral, una revisión sistemática. Fisioterapia. 2012; 34:225-34.
- [Background] Tseng SH, Chen HC, Tam KW. Systematic review and meta-analysis of the effect of equine assisted activities and therapies on gross motor outcome in children with cerebral palsy. Disabil Rehabil. 2013 Jan;35(2):89-99. doi: 10.3109/09638288.2012.687033. Epub 2012 May 26. PMID 22630812
- [Background] Martin-Valero R, Vega-Ballon J, Perez-Cabezas V. Benefits of hippotherapy in children with cerebral palsy: A narrative review. Eur J Paediatr Neurol. 2018 Nov;22(6):1150-1160. doi: 10.1016/j.ejpn.2018.07.002. Epub 2018 Jul 10. PMID 30017618
- [Background] Dewar R, Love S, Johnston LM. Exercise interventions improve postural control in children with cerebral palsy: a systematic review. Dev Med Child Neurol. 2015 Jun;57(6):504-20. doi: 10.1111/dmcn.12660. Epub 2014 Dec 18. PMID 25523410
- [Background] Mutoh T, Mutoh T, Takada M, Doumura M, Ihara M, Taki Y, Tsubone H, Ihara M. Application of a tri-axial accelerometry-based portable motion recorder for the quantitative assessment of hippotherapy in children and adolescents with cerebral palsy. J Phys Ther Sci. 2016 Oct;28(10):2970-2974. doi: 10.1589/jpts.28.2970. Epub 2016 Oct 28. PMID 27821971
- [Background] Mutoh T, Mutoh T, Tsubone H, Takada M, Doumura M, Ihara M, Shimomura H, Taki Y, Ihara M. Impact of serial gait analyses on long-term outcome of hippotherapy in children and adolescents with cerebral palsy. Complement Ther Clin Pract. 2018 Feb;30:19-23. doi: 10.1016/j.ctcp.2017.11.003. Epub 2017 Nov 8. PMID 29389473
- [Background] Matusiak-Wieczorek E, Malachowska-Sobieska M, Synder M. Influence of Hippotherapy on Body Balance in the Sitting Position Among Children with Cerebral Palsy. Ortop Traumatol Rehabil. 2016 Mar 23;18(2):165-175. doi: 10.5604/15093492.1205024. PMID 28155825
- [Background] Rigby BR, Gloeckner AR, Sessums S, Lanning BA, Grandjean PW. Changes in Cardiorespiratory Responses and Kinematics With Hippotherapy in Youth With and Without Cerebral Palsy. Res Q Exerc Sport. 2017 Mar;88(1):26-35. doi: 10.1080/02701367.2016.1266458. Epub 2017 Jan 11. PMID 28075704
- [Background] Strashko EY, Kapustianska capital A, CyrillicA, Bobyreva LE. Experience of using hippotherapy in complex effects on muscle spirals in children with spastic forms of cerebral palsy. Wiad Lek. 2016;69(3 pt 2):527-529. PMID 27717938
- [Background] Champagne D, Corriveau H, Dugas C. Effect of Hippotherapy on Motor Proficiency and Function in Children with Cerebral Palsy Who Walk. Phys Occup Ther Pediatr. 2017 Feb;37(1):51-63. doi: 10.3109/01942638.2015.1129386. Epub 2016 Mar 1. PMID 26930110
- [Background] Angsupaisal M, Visser B, Alkema A, Meinsma-van der Tuin M, Maathuis CG, Reinders-Messelink H, Hadders-Algra M. Therapist-Designed Adaptive Riding in Children With Cerebral Palsy: Results of a Feasibility Study. Phys Ther. 2015 Aug;95(8):1151-62. doi: 10.2522/ptj.20140146. Epub 2015 Apr 23. PMID 25908525
- [Background] De Miguel A, De Miguel MD, Lucena-Anton D, Rubio MD. [Effects of hypotherapy on the motor function of persons with Down's syndrome: a systematic review]. Rev Neurol. 2018 Oct 1;67(7):233-241. Spanish. PMID 30232796
- [Background] Kwon JY, Chang HJ, Yi SH, Lee JY, Shin HY, Kim YH. Effect of hippotherapy on gross motor function in children with cerebral palsy: a randomized controlled trial. J Altern Complement Med. 2015 Jan;21(1):15-21. doi: 10.1089/acm.2014.0021. Epub 2014 Dec 31. PMID 25551626
- [Background] Hsieh YL, Yang CC, Sun SH, Chan SY, Wang TH, Luo HJ. Effects of hippotherapy on body functions, activities and participation in children with cerebral palsy based on ICF-CY assessments. Disabil Rehabil. 2017 Aug;39(17):1703-1713. doi: 10.1080/09638288.2016.1207108. Epub 2016 Jul 20. PMID 27440177
- [Background] Lucena-Anton D, Rosety-Rodriguez I, Moral-Munoz JA. Effects of a hippotherapy intervention on muscle spasticity in children with cerebral palsy: A randomized controlled trial. Complement Ther Clin Pract. 2018 May;31:188-192. doi: 10.1016/j.ctcp.2018.02.013. Epub 2018 Feb 19. PMID 29705454
- [Background] Ribeiro MF, Espindula AP, Lage JB, Bevilacqua Junior DE, Diniz LH, Mello EC, Ferreira AA, Ferraz MLF, Teixeira VPA. Analysis of the electromiographic activity of lower limb and motor function in hippotherapy practitioners with cerebral palsy. J Bodyw Mov Ther. 2019 Jan;23(1):39-47. doi: 10.1016/j.jbmt.2017.12.007. Epub 2017 Dec 9. PMID 30691759
- [Background] Zaliene L, Mockeviciene D, Kreiviniene B, Razbadauskas A, Kleiva Z, Kirkutis A. Short-Term and Long-Term Effects of Riding for Children with Cerebral Palsy Gross Motor Functions. Biomed Res Int. 2018 Jul 8;2018:4190249. doi: 10.1155/2018/4190249. eCollection 2018. PMID 30069468
- [Background] Trzmiel T, Purandare B, Michalak M, Zasadzka E, Pawlaczyk M. Equine assisted activities and therapies in children with autism spectrum disorder: A systematic review and a meta-analysis. Complement Ther Med. 2019 Feb;42:104-113. doi: 10.1016/j.ctim.2018.11.004. Epub 2018 Nov 5. PMID 30670226
- [Background] Harris A, Williams JM. The Impact of a Horse Riding Intervention on the Social Functioning of Children with Autism Spectrum Disorder. Int J Environ Res Public Health. 2017 Jul 14;14(7):776. doi: 10.3390/ijerph14070776. PMID 28708075
- [Background] Llambias C, Magill-Evans J, Smith V, Warren S. Equine-Assisted Occupational Therapy: Increasing Engagement for Children With Autism Spectrum Disorder. Am J Occup Ther. 2016 Nov/Dec;70(6):7006220040p1-7006220040p9. doi: 10.5014/ajot.2016.020701. PMID 27767943
- [Background] Anderson S, Meints K. Brief Report: The Effects of Equine-Assisted Activities on the Social Functioning in Children and Adolescents with Autism Spectrum Disorder. J Autism Dev Disord. 2016 Oct;46(10):3344-52. doi: 10.1007/s10803-016-2869-3. PMID 27457363
- [Background] Borgi M, Loliva D, Cerino S, Chiarotti F, Venerosi A, Bramini M, Nonnis E, Marcelli M, Vinti C, De Santis C, Bisacco F, Fagerlie M, Frascarelli M, Cirulli F. Effectiveness of a Standardized Equine-Assisted Therapy Program for Children with Autism Spectrum Disorder. J Autism Dev Disord. 2016 Jan;46(1):1-9. doi: 10.1007/s10803-015-2530-6. PMID 26210515
- [Background] Ward SC, Whalon K, Rusnak K, Wendell K, Paschall N. The association between therapeutic horseback riding and the social communication and sensory reactions of children with autism. J Autism Dev Disord. 2013 Sep;43(9):2190-8. doi: 10.1007/s10803-013-1773-3. PMID 23371511
- [Background] Srinivasan SM, Cavagnino DT, Bhat AN. Effects of Equine Therapy on Individuals with Autism Spectrum Disorder: A Systematic Review. Rev J Autism Dev Disord. 2018 Jun;5(2):156-175. doi: 10.1007/s40489-018-0130-z. Epub 2018 Feb 20. PMID 30319932
- [Background] Tan VX, Simmonds JG. Parent Perceptions of Psychosocial Outcomes of Equine-Assisted Interventions for Children with Autism Spectrum Disorder. J Autism Dev Disord. 2018 Mar;48(3):759-769. doi: 10.1007/s10803-017-3399-3. PMID 29196865
- [Background] Garcia-Gomez A, Rodriguez-Jimenez M, Guerrero-Barona E, Rubio-Jimenez JC, Garcia-Pena I, Moreno-Manso JM. Benefits of an experimental program of equestrian therapy for children with ADHD. Res Dev Disabil. 2016 Dec;59:176-185. doi: 10.1016/j.ridd.2016.09.003. Epub 2016 Sep 7. PMID 27614276
- [Background] Hyun GJ, Jung TW, Park JH, Kang KD, Kim SM, Son YD, Cheong JH, Kim BN, Han DH. Changes in Gait Balance and Brain Connectivity in Response to Equine-Assisted Activity and Training in Children with Attention Deficit Hyperactivity Disorder. J Altern Complement Med. 2016 Apr;22(4):286-93. doi: 10.1089/acm.2015.0299. Epub 2016 Mar 16. PMID 26982567
- [Background] Oh Y, Joung YS, Jang B, Yoo JH, Song J, Kim J, Kim K, Kim S, Lee J, Shin HY, Kwon JY, Kim YH, Jeong B. Efficacy of Hippotherapy Versus Pharmacotherapy in Attention-Deficit/Hyperactivity Disorder: A Randomized Clinical Trial. J Altern Complement Med. 2018 May;24(5):463-471. doi: 10.1089/acm.2017.0358. Epub 2018 Apr 11. PMID 29641212
- [Background] Munoz-Lasa S, Lopez de Silanes C, Atin-Arratibel MA, Bravo-Llatas C, Pastor-Jimeno S, Maximo-Bocanegra N. Effects of hippotherapy in multiple sclerosis: pilot study on quality of life, spasticity, gait, pelvic floor, depression and fatigue. Med Clin (Barc). 2019 Jan 18;152(2):55-58. doi: 10.1016/j.medcli.2018.02.015. Epub 2018 Apr 19. English, Spanish. PMID 29680460
- [Background] Vermohlen V, Schiller P, Schickendantz S, Drache M, Hussack S, Gerber-Grote A, Pohlau D. Hippotherapy for patients with multiple sclerosis: A multicenter randomized controlled trial (MS-HIPPO). Mult Scler. 2018 Sep;24(10):1375-1382. doi: 10.1177/1352458517721354. Epub 2017 Aug 3. PMID 28770664
- [Background] Erdman EA, Pierce SR. Use of Hippotherapy With a Boy After Traumatic Brain Injury: A Case Study. Pediatr Phys Ther. 2016 Spring;28(1):109-16. doi: 10.1097/PEP.0000000000000204. PMID 27088700
- [Background] Cabiddu R, Borghi-Silva A, Trimer R, Trimer V, Ricci PA, Italiano Monteiro C, Camargo Magalhaes Maniglia M, Silva Pereira AM, Rodrigues das Chagas G, Carvalho EM. Hippotherapy acute impact on heart rate variability non-linear dynamics in neurological disorders. Physiol Behav. 2016 May 15;159:88-94. doi: 10.1016/j.physbeh.2016.03.012. Epub 2016 Mar 15. PMID 26988283
- [Background] Del Rosario-Montejo O, Molina-Rueda F, Munoz-Lasa S, Alguacil-Diego IM. Effectiveness of equine therapy in children with psychomotor impairment. Neurologia. 2015 Sep;30(7):425-32. doi: 10.1016/j.nrl.2013.12.023. Epub 2014 Mar 20. English, Spanish. PMID 24656851
- [Background] Hession CE, Eastwood B, Watterson D, Lehane CM, Oxley N, Murphy BA. Therapeutic horse riding improves cognition, mood arousal, and ambulation in children with dyspraxia. J Altern Complement Med. 2014 Jan;20(1):19-23. doi: 10.1089/acm.2013.0207. Epub 2013 Oct 2. PMID 24088010
- [Background] Kraft KA, Weisberg J, Finch MD, Nickel A, Griffin KH, Barnes TL. Hippotherapy in Rehabilitation Care for Children With Neurological Impairments and Developmental Delays: A Case Series. Pediatr Phys Ther. 2019 Jan;31(1):E14-E21. doi: 10.1097/PEP.0000000000000567. PMID 30557295
- [Background] Hession CE, Law Smith MJ, Watterson D, Oxley N, Murphy BA. The Impact of Equine Therapy and an Audio-Visual Approach Emphasizing Rhythm and Beat Perception in Children with Developmental Coordination Disorder. J Altern Complement Med. 2019 May;25(5):535-541. doi: 10.1089/acm.2017.0242. Epub 2019 Feb 21. PMID 30789282
- [Background] Wilson K, Buultjens M, Monfries M, Karimi L. Equine-Assisted Psychotherapy for adolescents experiencing depression and/or anxiety: A therapist's perspective. Clin Child Psychol Psychiatry. 2017 Jan;22(1):16-33. doi: 10.1177/1359104515572379. Epub 2016 Jul 27. PMID 26668260
- [Background] Alfonso SV, Alfonso LA, Llabre MM, Fernandez MI. Project Stride: An Equine-Assisted Intervention to Reduce Symptoms of Social Anxiety in Young Women. Explore (NY). 2015 Nov-Dec;11(6):461-7. doi: 10.1016/j.explore.2015.08.003. Epub 2015 Aug 20. PMID 26386749
- [Background] Frederick KE, Ivey Hatz J, Lanning B. Not Just Horsing Around: The Impact of Equine-Assisted Learning on Levels of Hope and Depression in At-Risk Adolescents. Community Ment Health J. 2015 Oct;51(7):809-17. doi: 10.1007/s10597-015-9836-x. Epub 2015 Feb 20. PMID 25698076
- [Background] Dezutti JE. Eating disorders and equine therapy: a nurse's perspective on connecting through the recovery process. J Psychosoc Nurs Ment Health Serv. 2013 Sep;51(9):24-31. doi: 10.3928/02793695-20130612-01. Epub 2013 Jun 21. PMID 23786240
- [Background] Rodriguez-Mansilla J, Gonzalez-Sanchez B, Torres-Piles S, Martin JG, Jimenez-Palomares M, Bellino MN. Effects of the application of therapeutic massage in children with cancer: a systematic review. Rev Lat Am Enfermagem. 2017 Jun 8;25:e2903. doi: 10.1590/1518-8345.1774.2903. PMID 28614430
- [Background] Capdevila L, Rodas G, Ocaña M, Parrado E, Pintanel M, Valero M. Heart rate variability as a health inicator in sports: validation with a health-related qualify of questionnaire (Short form-12). Apunts Medicina de l'Esport 2008; 43: 62-9.
- [Background] Heart rate variability. Standards of measurement, physiological interpretation, and clinical use. Task Force of the European Society of Cardiology and the North American Society of Pacing and Electrophysiology. Eur Heart J. 1996 Mar;17(3):354-81. No abstract available. PMID 8737210